CLINICAL TRIAL: NCT00838669
Title: Evaluation of the Effect of Food and Posture on the Pharmacokinetics of Paliperidone After a Single Administration of 12 mg ER OROS Paliperidone to Healthy Men
Brief Title: A Study of the Effect of Food and Posture on the Pharmacokinetics of a Single Dose of ER OROS Paliperidone
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CR006223
Record Dates: First submitted 2009-02-05; First posted 2009-02-06 (Estimated); Last update posted 2011-05-18 (Estimated); Status verified 2010-03

CONDITIONS: Schizophrenia
Keywords: Schizophrenia; Mood disorders; Antipsychotic drugs; Extended release OROS paliperidone
MeSH Terms: conditions — Schizophrenia; Mood Disorders

INTERVENTIONS:
Drug: Extended release OROS paliperidone

SUMMARY:
The purposes of this study are to evaluate the effect of food on the pharmacokinetics of extended-release (ER) OROS paliperidone in healthy men, and to evaluate the effect of posture on the pharmacokinetics of ER OROS paliperidone under fasting conditions. Additionally, the safety and tolerability of the treatments in healthy men will be assessed.

DETAILED DESCRIPTION:
The current study was designed to evaluate the effect of food on the pharmacokinetics of the to be marketed formulation of ER OROS paliperidone in mobile healthy men, which represents the normal conditions. The 12-mg ER OROS paliperidone ER by oral administration single dose used in this study does not require prolonged bed rest as a precautionary measure to prevent orthostatic hypotension. To support an evaluation of the effect of posture on the pharmacokinetics of ER OROS paliperidone under fasting conditions, study medication was also administered to healthy men in the fasted state while confined to bed for approximately 36 hours. The safety and tolerability of the treatments in healthy men will be assessed. 12 mg ER OROS paliperidone ER, oral administration, single dose

ELIGIBILITY:
Inclusion Criteria:

* Body mass index (weight [kg]/height [m2]) of 18 to 30 kg/m2, inclusive
* A supine (after 5 minutes rest) blood pressure between 100 and 140 mmHg systolic, inclusive, and 50 and 90 mmHg diastolic, inclusive
* Healthy on the basis of a prestudy physical examination, medical history, 12-lead ECG, and the laboratory results of serum chemistry, hematology, and urinalysis performed within 21 days before the first dose. If the results of the serum chemistry, hematology, or urinalysis testing are not within the laboratory's reference ranges, the male volunteer can be included only if the investigator judges that the deviations are not clinically significant. For renal function tests, the values must be within the normal laboratory reference ranges.

Exclusion Criteria:

* Known drug allergy to risperidone, paliperidone, or any of its excipients
* Known history of drug-induced dystonia
* Known allergy or history of significant hypersensitivity to heparin, if a heparin lock will be used
* Recent history of alcohol or substance abuse, a positive test result for the urine drug screen at screening or upon admittance to the testing facility, a positive result for the alcohol urine test upon admittance to the testing facility
* Relevant history or presence of any cardiovascular (including myocardial infarct or cardiac arrhythmia), respiratory, neurologic (including seizures), psychiatric, renal, hepatic, gastrointestinal (including surgeries, severe gastrointestinal narrowing, and malabsorption problems), endocrine, hematologic, or immunologic disease
* History of any cancer, with the exception of basal cell carcinomas
* History of smoking or use of nicotine-containing substances within the last 2 months, as determined by medical history and/or volunteer's verbal report. Volunteers must agree to refrain from use throughout the study

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 74 (Actual)
Dates: Start 2005-08; Study Completion 2005-12 (Actual)

PRIMARY OUTCOMES:
to evaluate the effect of food on the pharmacokinetics of ER OROS paliperidone in ambulant healthy men; to evaluate the effect of posture on the pharmacokinetics of ER OROS paliperidone under fasting conditions

SECONDARY OUTCOMES:
to evaluate the safety and tolerability of the treatments in healthy men

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Pharmaceutical Research & Development, L.L. C. Clinical Trial, Study Director — Johnson & Johnson Pharmaceutical Research & Development, L.L.C.

REFERENCES:
- See also: A study of the effect of food and posture on the pharmacokinetics of a single dose of ER OROS paliperidone — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=710&filename=CR006223_CSR.pdf